CLINICAL TRIAL: NCT05307328
Title: SPI-62 as a Treatment for Adrenocorticotropic Hormone-dependent Cushing's Syndrome
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sparrow Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPI-62-CL-2001
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-05

CONDITIONS: Cushing's Syndrome I; Cushing Disease Due to Increased ACTH Secretion; Cortisol Excess; Cortisol; Hypersecretion; Cortisol Overproduction; Ectopic ACTH Secretion
Keywords: Cushing's Syndrome; ACTH Secretion; Cushing's Disease; Excessive Cortisol secretion; Cortisol; ectopic CRH secretion
MeSH Terms: conditions — ACTH Syndrome, Ectopic; Cushing Syndrome; Pituitary ACTH Hypersecretion

STUDY DESIGN:
Intervention Model Description: Staggered parallel crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- SPI-62 (Experimental): Active drug by mouth each morning for up to 12 weeks
  Interventions: Drug: SPI-62; Drug: Placebo
- Placebo (Placebo Comparator): Placebo by mouth each morning for up to 12 weeks
  Interventions: Drug: SPI-62; Drug: Placebo

INTERVENTIONS:
Drug: SPI-62 — 11β hydroxysteroid dehydrogenase type 1 (HSD-1) inhibitor
Drug: Placebo — Inactive tablets identical to SPI-62 tablets

SUMMARY:
This is a randomized, placebo-controlled, study of SPI-62 in subjects with ACTH-dependent Cushing's syndrome caused by a non-adrenal tumor. Subjects will receive each of the following 2 treatments for 24 weeks: SPI-62 and matching placebo with the option of long-term extension.

DETAILED DESCRIPTION:
This is a multicenter, randomized, placebo-controlled, Phase 2 study to evaluate the pharmacologic effect, efficacy, and safety of SPI-62 in subjects with ACTH-dependent Cushing's syndrome. Each subject who provides consent and meets all inclusion and exclusion criteria will participate in a screening period (Days -35 to -8), a baseline period (Days -7 to -1), and a treatment period (Day 1 of Week 1 to Day 168 ± 3 days of Week 24) and, the option of long-term extension. Subjects have the option to continue with the study on active study drug and return to the site every 3 months for blood tests and study drug dispensing. The visits may be conducted remotely if testing can be arranged.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-menstruating female
* 18 years or older
* Active and consistent cortisol excess
* Documented diagnosis of ACTH-dependent Cushing's syndrome including Cushing's disease, ectopic ACTH secretion, and ectopic CRH secretion.

Exclusion Criteria:

* Recent (within 6 weeks) surgery for Cushing's or surgery planned within 24 weeks of randomization.
* History of any fractionated radiation therapy for Cushing's within the past 2 years or conventional radiation therapy within 4 years.
* History of bilateral adrenalectomy or exogenous, pseudo, cyclic, or non-ACTH-dependent Cushing's syndrome (including certain inherited conditions).
* High risk of acute morbidity from corticotroph adenoma growth (similar to that which occurs with Nelson's syndrome) defined as current evidence of macroadenoma at risk of impingement of vital structures.
* Any current or prior medical condition, medical or surgical therapies, or clinical trial participation expected to interfere with the conduct of the study or the evaluation of its results, including but not limited to poor venous access or recent receipt or donation of blood products.
* Women who are currently pregnant, lactating or planning fertility and unwilling to adhere to approved contraceptives or abstinence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urinary HSD-1 ratio | Baseline to 6 weeks
  The urinary HSD-1 ratio (tetrahydrocortisol + allotetrahydrocortisol ) / tetrahydrocortisone will be used as a biomarker of HSD-1 activity in liver. The primary analysis will include only subjects with Cushing's disease.

SECONDARY OUTCOMES:
Treatment emergent adverse events | Baseline through 24 weeks of treatment
  Adverse events including clinically significant abnormal values on clinical laboratory evaluations, continuous glucose monitoring (CGM), 12-lead ECGs, vital signs measurements (including orthostatic vital sign measurements), physical examinations, and HPA and HPG axis biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Frank Czerwiec, MD, Study Director — Sparrow Pharmaceuticals (info@sparrowpharma.com)
Locations (12):
- United States (8):
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Institute (BNI) - Pituitary Center, Phoenix, Arizona
  - Southwest General Healthcare Center, Fort Myers, Florida
  - Mayo Clinic Cancer Center (MCCC) - Rochester, Rochester, Minnesota
  - Washington University School of Medicine - Center for Advanced Medicine (CAM), St Louis, Missouri
  - Comprehensive and Interventional Pain Management Llp, Henderson, Nevada
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oregon Health & Science University (OHSU) - Northwest Pituitary Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
- Bulgaria (3):
  - Medical University of Plovdiv, Plovdiv
  - Clinical Center of Endocrinology and Gerontology, University Hospital of Endocrinology, Medical University Sofia (USHATE), Sofia
  - Medical University of Sofia, Sofia
- Carol Davila University of Medicine and Pharmacy, Bucharest, Romania